CLINICAL TRIAL: NCT06318741
Title: Effects of Aerobic Exercise on Kinesiophobia, Functional Capacity and Quality of Life in Obese Patients with Atherosclerotic Cardiovascular Disease
Brief Title: Effects of Aerobic Exercise in Obese Patients with Atherosclerotic Cardiovascular Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, Professor Doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KayseriCHkinezyofobi
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Coronary Artery Disease
MeSH Terms: conditions — Obesity; Coronary Artery Disease | interventions — Posture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hospital exercise group (Active Comparator): According to the Cardiopulmonary exercise test (KPET) test in Group 1 (medium intensity continuous exercise group), 50 minutes (5 minutes warm-up, 40 minutes exercise, 5 minutes exercise, 5 minutes warm-up, 40 minutes exercise, 5 minutes) for 8 weeks, 3 days a week, at an exercise intensity of 50-60% of the VO2 max level recorded individually in the patients. Aerobic exercise therapy will be organized to be applied on a treadmill (in the form of a minute cool-down).
  Interventions: Other: aerobic exercise on the treadmill+For both groups, patients will be recommended joint range of motion (ROM), stretching, strengthening, posture and balance and flexibility exercises for all joints.
- home exercise group (Placebo Comparator): For the home exercise group, walking for 50 minutes, 3 days a week, with an intensity of 12-13 Rate of perceived exertion (RPE) according to the Modified Borg scale will be recommended for 8 weeks.
  Interventions: Other: Walking at an intensity of 12-13 RPE+For both groups, patients will be recommended ROM, stretching, strengthening, posture and balance and flexibility exercises for all joints.

INTERVENTIONS:
Other: aerobic exercise on the treadmill+For both groups, patients will be recommended joint range of motion (ROM), stretching, strengthening, posture and balance and flexibility exercises for all joints. — aerobic exercise on the treadmill
  Arms: hospital exercise group
Other: Walking at an intensity of 12-13 RPE+For both groups, patients will be recommended ROM, stretching, strengthening, posture and balance and flexibility exercises for all joints. — Walking at an intensity of 12-13 RPE
  Arms: home exercise group

SUMMARY:
Obesity is classified using body mass index (BMI) (BMI ≥25 overweight, BMI ≥30 obese, BMI ≥40 morbidly obese). Obese patients are Class 1 according to BMI; BMI:30-34.9 and Class 2; BMI: It is classified as 35-39.9. Patients with classes 1 and 2 will be included in the study. Obesity can be accompanied by comorbidities such as atherosclerotic vascular and cardiac pathologies, hyperlipidemia, hypertension, coronary artery disease, diabetes mellitus, so obesity treatment should be managed multidisciplinary. The basic approach to obesity treatment is diet, exercise, medical treatment, treatment of comorbid conditions and surgery. Aerobic exercise therapy, which is one of the conservative approaches in the treatment of obesity, also has an important place in the treatment of cardiovascular diseases associated with obesity. Atherosclerotic cardiovascular disease (AKD) is one of the most important causes of morbidity and mortality worldwide. Negative changes in functional capacity, quality of life and psychosocial situations are observed due to disorders associated with this disease. Physical activity is among the modifiable risk factors in atherosclerotic diseases. However, patients have a fear of movement related to angina-like symptoms, with the thought that the symptoms may recur during exercise. Lack of physical activity due to fear of movement leads to obesity, which in turn leads to aggravation of atherosclerosis and an increase in the incidence of cardiovascular events, which negatively affects individual and psychosocial capacity. Cardiopulmonary exercise test (CPET) is a non-invasive procedure that evaluates the individual's capacity during dynamic exercise and provides diagnostic and prognostic information. CPET is based on the investigation of the respiratory system, cardiovascular system and cellular response to exercise performed under controlled metabolic conditions. It allows holistic evaluation of the response to exercise, including not only the pulmonary and cardiovascular systems but also the musculoskeletal system. Fear of movement or kinesiophobia; It is defined as a state of fear and avoidance of activity and physical movement resulting from the feeling of sensitivity to painful injury and repeated injury.

DETAILED DESCRIPTION:
Obesity, defined by the World Health Organization (WHO) as "abnormal or excessive fat accumulation in the body that negatively affects health", has become an important public health problem that affects the quality of life at individual and social levels. Obesity is defined by using body mass index (BMI) (BMI ≥ 25 patients are classified as overweight, BMI ≥30 as obese, BMI ≥40 as morbidly obese. Obese patients are classified according to BMI as Class 1, BMI: 30-34.9 and Class 2, BMI: 35-39.9. Class 1 and 2 patients were included in the study. Patients will be included. Obesity can be accompanied by comorbidities such as atherosclerotic vascular and cardiac pathologies, hyperlipidemia, hypertension, coronary artery disease, diabetes mellitus and chronic musculoskeletal disorders such as osteoarthritis, low back pain and fibromyalgia. Therefore, obesity treatment should be managed multidisciplinary. The basic approach in obesity treatment is diet. , exercise, medical treatment, treatment of comorbid conditions and surgery.Aerobic exercise therapy, which is one of the conservative approaches in the treatment of obesity, also has an important place in the treatment of cardiovascular diseases associated with obesity. Atherosclerotic cardiovascular disease (AKD) is one of the most important causes of morbidity and mortality worldwide. Negative changes in functional capacity, quality of life and psychosocial situations are observed due to disorders associated with this disease. Physical activity is among the modifiable risk factors in atherosclerotic diseases. However, patients have a fear of movement related to angina-like symptoms, with the thought that the symptoms may recur during exercise. Lack of physical activity due to fear of movement leads to obesity, which in turn leads to aggravation of atherosclerosis and an increase in the incidence of cardiovascular events, which negatively affects individual and psychosocial capacity. Anthropometry is the investigation of measurements of the human body in terms of bone dimensions, muscle and fat tissue. Anthropometric measurements are measurements that reveal the composition and body size / structure of the human body. Anthropometric measurements gain importance when evaluating the nutritional status of people because they show body fat storage and protein storage. Evaluation of growth and body composition, that is, body fat and lean body tissue, can be determined by anthropometric measurements. Anthropometric measurements help analyze the relationship between obesity and diseases. Anthropometric measurements are important for evaluating the nutritional status of a population or individual. Cardiopulmonary exercise test (CPET) is a non-invasive procedure that evaluates the individual's capacity during dynamic exercise and provides diagnostic and prognostic information. CPET is based on the investigation of the respiratory system, cardiovascular system and cellular response to exercise performed under controlled metabolic conditions. It allows holistic evaluation of the response to exercise, including not only the pulmonary and cardiovascular systems but also the musculoskeletal system. Fear of movement or kinesiophobia; It is defined as a state of fear and avoidance of activity and physical movement resulting from the feeling of sensitivity to painful injury and repeated injury. Kinesiophobia is assessed with the Tampa Kinesiophobia Scale. This scale, consisting of 17 items, evaluates how afraid patients are of moving their bodies. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement. Each item is scored on a 4-point Likert Scale; 1-4. The answers and their numerical values are as follows: 1; Strongly disagree, 2; disagree, 3; agree and 4; I totally agree. The scores of items 4, 8, 12 and 16 should be reversed when calculating the total score. The total score obtained by adding different items may vary between 17 and 68. Previous studies have shown that this scale is generally applied to patients with low back pain, knee osteoarthritis, lymphedema and osteoporosis. In the literature, there are limited age group and uncontrolled studies in patients with cardiovascular disease. However, to the best of this knowledge, this study will be one of the limited number of blind, prospective, randomized controlled studies in the literature that evaluate fear of movement in obese patients with atherosclerotic cardiovascular disease who receive aerobic exercise therapy. The aim of this study is to investigate the effects of an aerobic exercise program on anthropometric measurements, kinesiophobia, psychosocial status, physical activity level and quality of life in obese individuals with atherosclerotic cardiovascular disease. This hypothesis in this study is that an aerobic exercise program will cause significant changes in anthropometric measures, kinesiophobia and quality of life in obese patients with atherosclerotic heart disease. In this study, it is expected that a regular, supervised aerobic exercise program will create a more effective response in terms of physical, psychosocial and patient compliance in the individual compared to a home exercise program in obese individuals who often have a sedentary lifestyle, and therefore will provide a change in anthropometric measurements. Patients who are admitted to Kayseri City Hospital Physical Medicine and Rehabilitation Clinic Cardiopulmonary Rehabilitation Unit, between the ages of 18-65, with a BMI of 30-40, with class 1 and 2 obese atherosclerotic cardiovascular pathology, and with American Heart Association stage B and New York Heart Association class 1 will be included in this study. Patients participating in the study will be randomized into 2 groups: moderate-intensity continuous exercise group (Group 1) and home exercise group (Group 2). The change in the average Tampa Scale Kinesiophobia (TSK) score of each group over time will be evaluated within the 0th, 8th and 20th weeks. Additionally, the change in the average TSK scores between the two groups over time (0th, 8th and 20th weeks) will be compared. In this hypothesis; A decrease in TSK score is expected over time with the exercise program. The minimum sample size required to find a significant difference between both groups was determined by Jiménez et al. It was calculated in the G*Power 3.1.9.4 program, using the study as a reference. According to these criteria; While the power of the test (1-β) is 0.80, the amount of type-1 error (α) is 0.05, and the alternative hypothesis (H1) is one-sided, the minimum sample size required to find a significant difference between the groups is a total of 28 patients, 14 patients in each group. calculated as a patient. The dropout rate was estimated to be 10%. Therefore, a total of 32 patients will be included in the study, 16 patients in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Class 1 and class 2 obese patients with a BMI of 30 kg/m2 and above and below 40 kg/m2
2. Patients with atherosclerotic cardiovascular disease diagnosed by angiography
3. Women and men aged 18-65
4. Individuals who agree to participate in the study and have received a written voluntary consent form.

Exclusion Criteria:

1. Clinical neuromuscular diseases that limit exercise, previous diagnosis of asthma, congestive heart failure, unstable angina, uncontrolled psychiatric disease or cognitive-cognitive disorders (confirmed and diagnosed in International Classification of Disease (ICD)-10 diagnosis codes 'Schizophrenia and Psychotic states (F20, F20.0, F20.1, F20.2, F20.3, F20.4, F20.5, F20.6, F20.8, F20.9, F06.2, F23.0, F23.1, F23.2, F29) , Bipolar Disorder (F31, F31.0, F31.1, F31.2, F31.3, F31.4, F31.5, F31.6, F31.7, F31.8, F31.9) and Substance Abuse (Patients with diagnosis code ' (Z86.4)')
2. Presence of uncontrolled systemic diseases

   * Uncontrolled hypertension,
   * Uncontrolled diabetes mellitus,
   * Chronic liver failure
   * Chronic renal failure and dialysis patients
   * Chronic obstructive pulmonary disease and asthma
3. Malignancy
4. Infection
5. High fever
6. Acute inflammatory rheumatic diseases
7. Acute peripheral vascular diseases
8. Smoking before exercise test
9. Alcohol consumption before exercise test
10. Use of medications known to affect physical performance, heart rate or metabolism (including Beta blockers)
11. Patients without cooperation and compliance
12. Patients who did not agree to participate in the study
13. Patients who have been included in the cardiopulmonary rehabilitation (CPR) program in the last year
14. With acute coronary syndrome
15. Troponin positive
16. Unstable angina pectoris
17. Basic contraindications of exercise test:

    * High risk unstable angina
    * Acute Cardiac Diseases (Acute MI, Acute endocarditis, myocarditis or pericarditis, Acute pulmonary embolism, etc.)
    * Uncontrolled arrhythmias that can disrupt the hemodynamic response
    * Symptomatic severe aortic stenosis
    * Decompensated heart failure
    * Non-cardiac pathologies that will affect exercise performance and be aggravated by exercise (e.g. infection, renal failure, thyrotoxicosis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | week 0, 8th week, 20th week
  Fear of movement or kinesiophobia; It is defined as a state of fear and avoidance of activity and physical movement resulting from the feeling of sensitivity to painful injury and repeated injury. This scale, consisting of 17 items, evaluates how afraid patients are of moving their bodies. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement. Each item is scored on a 4-point Likert Scale.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test | week 0, 8th week, 20th week
  Cardiopulmonary exercise test (CPET) is a non-invasive procedure that evaluates the individual's capacity during dynamic exercise and provides diagnostic and prognostic information. CPET is based on the investigation of the respiratory system, cardiovascular system and cellular response to exercise performed under controlled metabolic conditions. It allows holistic evaluation of the response to exercise, including not only the pulmonary and cardiovascular systems but also the musculoskeletal system.
6 Minutes Walking Test | week 0, 8th week, 20th week
  It is a frequently used test in cardiopulmonary rehabilitation to monitor exercise capacity and treatment effectiveness. The patient should rest by sitting in a chair for 15 minutes before the test and wear appropriate shoes and comfortable clothing. Calculate the distance walked by the patient at their own walking pace in 6 minutes, preferably in a 30-meter long corridor.
Body anthropometric measurements | week 0, 8th week, 20th week
  Waist circumference, hip circumference, waist/hip ratio, waist/height ratio.
Hospital anxiety and depression scale | week 0, 8th week, 20th week
  The Hospital Anxiety and Depression (HADS) Scale was prepared to screen for anxiety and depression in people with physical illnesses.
international physical activity score | week 0, 8th week, 20th week
  It is a survey consisting of 7 questions that patients will answer and provides information about the time spent in sitting, walking, moderate and vigorous activities. The total score is obtained by calculating the time (minutes) and weekly frequencies (days) spent in these activities.
MacNew Heart Disease Health-Related Quality of Life Survey | week 0, 8th week, 20th week
  It is designed to assess the patient's feelings about how ischemic heart disease affects daily functioning and includes 27 items, a global HRQoL score and physical limitation, emotional, and social function subscales, along with a summary of available international results.
Numerical Rating Scale | week 0, 8th week, 20th week
  It is used as a measure of pain intensity in adults. 0;no pain, 10; It is the strongest pain felt

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gül Ülkü Demir, MD, Study Director — Kayseri City Hospital; Selim Oğuz, MD, Principal Investigator — Health Sciences University, Kayseri Medical Faculty
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apovian CM. Obesity: definition, comorbidities, causes, and burden. Am J Manag Care. 2016 Jun;22(7 Suppl):s176-85. PMID 27356115
- [Background] Jackson VM, Breen DM, Fortin JP, Liou A, Kuzmiski JB, Loomis AK, Rives ML, Shah B, Carpino PA. Latest approaches for the treatment of obesity. Expert Opin Drug Discov. 2015;10(8):825-39. doi: 10.1517/17460441.2015.1044966. Epub 2015 May 12. PMID 25967138
- [Background] Libby P, Theroux P. Pathophysiology of coronary artery disease. Circulation. 2005 Jun 28;111(25):3481-8. doi: 10.1161/CIRCULATIONAHA.105.537878. PMID 15983262
- [Background] Wood DW, Haig AJ, Yamakawa KS. Fear of movement/(re)injury and activity avoidance in persons with neurogenic versus vascular claudication. Spine J. 2012 Apr;12(4):292-300. doi: 10.1016/j.spinee.2012.02.015. Epub 2012 Apr 4. PMID 22480530
- [Background] Gazarova M, Galsneiderova M, Meciarova L. Obesity diagnosis and mortality risk based on a body shape index (ABSI) and other indices and anthropometric parameters in university students. Rocz Panstw Zakl Hig. 2019;70(3):267-275. doi: 10.32394/rpzh.2019.0077. PMID 31515986
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Weermeijer JD, Meulders A. Clinimetrics: Tampa Scale for Kinesiophobia. J Physiother. 2018 Apr;64(2):126. doi: 10.1016/j.jphys.2018.01.001. Epub 2018 Mar 19. No abstract available. PMID 29567379
- [Background] Cruz-Diaz D, Romeu M, Velasco-Gonzalez C, Martinez-Amat A, Hita-Contreras F. The effectiveness of 12 weeks of Pilates intervention on disability, pain and kinesiophobia in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 Sep;32(9):1249-1257. doi: 10.1177/0269215518768393. Epub 2018 Apr 13. PMID 29651872
- [Background] Areeudomwong P, Buttagat V. Reliability and Validity of the Cross-Culturally Adapted Thai Version of the Tampa Scale for Kinesiophobia in Knee Osteoarthritis Patients. Malays J Med Sci. 2017 Mar;24(2):61-67. doi: 10.21315/mjms2017.24.2.8. Epub 2017 Apr 14. PMID 28894405
- [Background] Gencay Can A, Can SS, Eksioglu E, Cakci FA. Is kinesiophobia associated with lymphedema, upper extremity function, and psychological morbidity in breast cancer survivors? Turk J Phys Med Rehabil. 2018 Aug 12;65(2):139-146. doi: 10.5606/tftrd.2019.2585. eCollection 2019 Jun. PMID 31453554
- [Background] Gunendi Z, Eker D, Tecer D, Karaoglan B, Ozyemisci-Taskiran O. Is the word "osteoporosis" a reason for kinesiophobia? Eur J Phys Rehabil Med. 2018 Oct;54(5):671-675. doi: 10.23736/S1973-9087.18.04931-6. Epub 2018 Feb 7. PMID 29422485
- [Background] Adachi H. Cardiopulmonary Exercise Test. Int Heart J. 2017 Oct 21;58(5):654-665. doi: 10.1536/ihj.17-264. Epub 2017 Sep 30. PMID 28966333
- [Background] Hamilton DM, Haennel RG. Validity and reliability of the 6-minute walk test in a cardiac rehabilitation population. J Cardiopulm Rehabil. 2000 May-Jun;20(3):156-64. doi: 10.1097/00008483-200005000-00003. PMID 10860197
- [Background] Sakamoto M, Suematsu Y, Yano Y, Kaino K, Teshima R, Matsuda T, Fujita M, Tazawa R, Fujimi K, Miura SI. Depression and Anxiety Are Associated with Physical Performance in Patients Undergoing Cardiac Rehabilitation: A Retrospective Observational Study. J Cardiovasc Dev Dis. 2022 Jan 11;9(1):21. doi: 10.3390/jcdd9010021. PMID 35050231
- [Background] Wang Y, Cao J, Kong X, Wang S, Meng L, Wang Y. The effects of CPET-guided cardiac rehabilitation on the cardiopulmonary function, the exercise endurance, and the NT-proBNP and hscTnT levels in CHF patients. Am J Transl Res. 2021 Jun 15;13(6):7104-7114. eCollection 2021. PMID 34306470
- [Background] Benetti M, Araujo CL, Santos RZ. Cardiorespiratory fitness and quality of life at different exercise intensities after myocardial infarction. Arq Bras Cardiol. 2010 Sep;95(3):399-404. doi: 10.1590/s0066-782x2010005000089. Epub 2010 Jul 16. PMID 20640381
- [Background] Verbrugghe J, Agten A, Stevens S, Hansen D, Demoulin C, O Eijnde B, Vandenabeele F, Timmermans A. Exercise Intensity Matters in Chronic Nonspecific Low Back Pain Rehabilitation. Med Sci Sports Exerc. 2019 Dec;51(12):2434-2442. doi: 10.1249/MSS.0000000000002078. PMID 31269004